CLINICAL TRIAL: NCT02130206
Title: The Microbiology of Caries Resistance. Subtitle: Functional Amyloid Formation in Streptococcus Mutans
Brief Title: The Microbiology of Caries Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 665-2008; A-2013-197-OC (Other: Colgate Palmolive)
Record Dates: First submitted 2014-04-25; First posted 2014-05-05 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Dental Caries
Keywords: Plaque, Saliva, Cavities
MeSH Terms: conditions — Dental Caries; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caries Free (Active Comparator): Gums will be examined. On some visits Saliva and plaque will be collected. Toothpaste assigned will include DenClude 1.5% Arginine.
  Interventions: Other: Caries Free
- Caries Free - Placebo (Placebo Comparator): Gums will be examined. On some visits Saliva and plaque will be collected. Marketed Toothpaste will be assigned.
  Interventions: Other: Caries Free - Placebo
- Caries Active (Active Comparator): Gums will be examined. On some visits Saliva and plaque will be collected. Toothpaste assigned will include DenClude 1.5% Arginine.
  Interventions: Other: Caries Active
- Caries Active - Placebo (Placebo Comparator): Gums will be examined. On some visits Saliva and plaque will be collected. Marketed Toothpaste will be assigned.
  Interventions: Other: Caries Active - Placebo

INTERVENTIONS:
Other: Caries Free — Gums will be examined. On some visits Saliva and plaque will be collected. Toothpaste assigned will include DenClude 1.5% Arginine.
  Arms: Caries Free
Other: Caries Active — Gums will be examined. On some visits Saliva and plaque will be collected. Toothpaste assigned will include DenClude 1.5% Arginine.
  Arms: Caries Active
Other: Caries Free - Placebo — Gums will be examined. On some visits Saliva and plaque will be collected. Marketed Toothpaste will be assigned.
  Arms: Caries Free - Placebo
Other: Caries Active - Placebo — Gums will be examined. On some visits Saliva and plaque will be collected. Marketed Toothpaste will be assigned.
  Arms: Caries Active - Placebo

SUMMARY:
The purpose of this research study is to investigate the bacterial composition of plaque and saliva located in the mouth and associate that with risk factors that cause cavities.

DETAILED DESCRIPTION:
Pre-Screening - If the subject chooses to be pre-screened for this study they will be asked to fill out a study registration form and an oral habits/medical history form. They will be asked to sign an Informed Consent. The subject will then have their teeth and gums examined. At this visit, the investigator will assess whether or not the subject is a good candidate for the study. During the phone interview each subject was asked not to brush or floss their teeth and not to eat or drink anything other than water for 8 hours prior to the pre-screening visit (Visit 0). If the subject was compliant with these requests, oral samples will be collected at this pre-screening visit and will now be considered Visit 1 (Baseline). If not, they will be asked to return to the clinic for another visit and asked not to brush or floss their teeth and not to eat or drink anything other than water 8 hours prior to that appointment. This visit will then be consider Visit 1 (Baseline).

Visit 1 (Baseline) - The subject will have their medical and dental history reviewed. They will have their teeth and gums examined. Saliva and plaque will be collected. Each subject will be given a toothbrush and toothpaste and instructed to not use any other dental products. This will be considered the "washout" period.

Visit 2 - The subject will be asked to return the unused toothpaste. Their medical and dental history will be reviewed and they will have their teeth examined. Saliva and plaque will be collected at this visit. The subjects will then be randomly assigned (by chance, like the flip of a coin) to the group that will use a marketed fluoride-containing toothpaste or to the group that will use a marketed arginine containing toothpaste. The subject will also be instructed not to brush or floss their teeth or eat or drink anything other than water for 8 hours prior to your next appointment.

Visits 3, 4, and 5 - Subjects will not be allowed to brush or floss their teeth or eat or drink anything other than water 8 hours prior to these visits. Saliva and plaque will be collected. On the 5th visit subjects will be asked to return the unused toothpaste tube. At this time participation in this research study will end and they will be instructed to return to their regular oral hygiene regiments.

ELIGIBILITY:
Inclusion Criteria:

* Twenty natural teeth excluding third molars
* No contraindications to dental treatment
* Caries Free
* Caries Active (at least two active sites)

Exclusion Criteria:

* Less that twenty teeth
* Any systemic disease that can cause xerostomia
* Taking medications that cause xerostomia
* Antibiotics last three months
* Advanced Periodontal Disease
* Removable or fixed dental appliances
* Bleeding disorders or taking anticoagulant medications
* Immune compromised individuals
* Participating in another research study
* Used flavored products such as mint flavored candies and chewing gum one week prior to or during the study
* Uses tobacco products
* Unwilling or unable to provide Informed Consent and follow collection instructions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from baseline to month 2 | Changes from baseline to month 2 (Screening)
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from month 2 to week 4 | Changes from month 2 to week 4 (Baseline)
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from week 4 to week 2 | Changes from week 4 to week 2 (Washout)
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from week 2 to week 8 | Changes from week 2 to week 8 (Evaluation)
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from week 8 to week 12 | Changes from week 8 to week 12 (Evaluation)
  Saliva and dental plaque will be collected during the study visit. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured using a standardized protocol.

SECONDARY OUTCOMES:
Bacteria collected from oral samples of healthy and caries-active subjects changes from baseline to month 2 | Changes from baseline to month 2 (Screening)
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects changes from month 2 to week 4 | Changes from month 2 to week 4 (Baseline)
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects changes from week 4 to week 2 | Changes from week 4 to week 2 (Washout)
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects changes from week 2 to week 8 | Changes from week 2 to week 8 (Evaluation)
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.
Bacteria collected from oral samples of healthy and caries-active subjects changes from week 8 to week 12 | Changes from week 8 to week 12 (Evaluation)
  Saliva and dental plaque will be collected during the baseline study visit. These oral samples will be plated in specific medium for bacterial growth and isolation. The isolated bacteria will be identified by molecular and microbiological techniques to characterize their capacity to produce ammonia from arginine - ADS activity. Protocols will be used to determine the sensitivity of the ADS of the oral isolates to environmental oral factors.

OTHER OUTCOMES:
Salivary factors present in healthy and caries-active subjects during the research study. | Up to six months.
  Saliva will be collected from healthy and caries-active subjects during the research study. Microbiological and molecular techniques such as microscopic observation of green birefringence, elisa assays and microRNA analysis will be used to determine and compare differences between salivary factors present in these two groups

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Nascimento, DDS, MS, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Dentistry, Gainesville, Florida, United States